CLINICAL TRIAL: NCT03305237
Title: The Big Breakfast Study: Chrono-nutrition Influence on Energy Expenditure and Body Weight
Brief Title: The Meal Time Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Collaborators: University of Surrey (Other); Maastricht University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 806; MR/P012205/1 (Other Grant/Funding Number: Medical Research Council)
Record Dates: First submitted 2017-09-26; First posted 2017-10-09 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Obesity; Weight Loss
Keywords: Weight loss; Chrono-nutrition; Diet; energy expenditure
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- big breakfast (BB) to big dinner (BD) (Experimental): Phase 1: no intervention, habitual diet for 4 days and then 4day maintenance diet Phase 2: consumption of BB energy restriction diets for 4 weeks Phase 3: washout for 1 week, controlled maintenance diet Phase 4: consumption of BD energy restriction diets for 4 weeks
  Interventions: Other: Big Breakfast; Other: Big Dinner
- big dinner (BD) to big breakfast (BB) (Experimental): Phase 1: no intervention, habitual diet for 4 days and then 4day maintenance diet Phase 2: consumption of BD energy restriction diets for 4 weeks Phase 3: washout for 1 week, controlled maintenance diet Phase 4: consumption of BB energy restriction diets for 4 weeks
  Interventions: Other: Big Breakfast; Other: Big Dinner

INTERVENTIONS:
Other: Big Breakfast — Weight loss diet (Calories fed to measured RMR) with calories distributed predominantly at breakfast (percent daily calories split between breakfast, lunch and dinner as 45-35-20%). The diet will be high protein (30% protein, 35% fat and 35% CHO) with all meals provided.
Other: Big Dinner — Weight loss diet (Calories fed to measured RMR) with calories distributed predominantly at dinner (percent daily calories split between breakfast, lunch and dinner as 20-35-45%). The diet will be high protein (30% protein, 35% fat and 35% CHO) with all meals provided.

SUMMARY:
This weight loss study will investigate the impact of calorie distribution across a day (large breakfast meals and smaller evening meals versus small breakfast meals and large evening meals) on body weight, and physiological and behavioral mechanisms regulating energy balance.

Participants will undergo 2 x 4 week energy restriction protocols in a randomized cross over design; big breakfast (45% of calories in the morning meal, 20% at dinner) and big dinner (45% of calories in the evening meal, 20% at breakfast). We predict that timing of eating will influence energy balance, because morning energy expenditure is amplified in comparison to the evening. This study will allow us to assess whether the increased energy expenditure in the morning is linked to natural biological circadian rhythm or behavioral adaptions.

DETAILED DESCRIPTION:
Dietary advice for weight management is broadly based on the assumption that a 'calorie is a calorie' and it does not matter when calories are consumed across the day. Recent evidence has challenged this assumption, suggesting that we may utilize calories more efficiently when consumed in the morning relative to the evening, and this could be used as a beneficial strategy for weight loss - this is a newly developing field of investigation which merges circadian biology with nutrition (chrono-nutrition).

Timing of food consumption is a modifiable factor influencing energy balance and body weight (and thus, disease risk). Previous research has shown that calories ingested at different times of the day have different effects on energy utilization, leading to differential weight loss, even at iso-caloric amounts. This study will aim to increase our understanding of the underlying behavioral and physiological mechanisms associated with differential weight loss and energy balance when calories are consumed predominantly in the morning versus in the evening.

This study will be a cross-over study comparing large breakfast versus large evening meals (percent daily calories split between breakfast, lunch and dinner as 45-35-20 (breakfast-loaded) or 20-35-45 (evening-loaded)) during energy restriction (Fed to measured RMR) on energy balance, through differences in both physiological and behavioural changes in energy expenditure and substrate utilization.

ELIGIBILITY:
Inclusion Criteria:

* BMI ranging from 27-42 kg/m2;
* Those habitually consuming breakfast (at least 5 times a week).

Exclusion Criteria:

* women who are pregnant, planning to be pregnant or breastfeeding
* subjects with food allergies which prevent consumption of the study diet.
* diagnosis of diabetes, hypertension, renal, hepatic, haematological disease, coronary heart disease, metabolic disease, gastrointestinal disease
* having given a pint of blood for transfusion purposes within the last month
* unsuitable veins for blood sampling
* inability to understand the participant information sheet
* inability to speak, read and understand the English language
* those on any prescription medications (other than oral contraceptives) which will adversely affect the study outcomes (i.e. medications affecting, circadian timing, sleep or metabolic function).
* those on any specific diet regimes
* those on any weight loss programmes (that may be affecting lifestyle, physical activity and diet).
* Extremes of chronotypes, sleep patterns and physical activity.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Energy balance | Measured up to day 71 of study
  Change in energy balance during each diet protocol (body weight (kg))

SECONDARY OUTCOMES:
Total Daily Energy Expenditure | 4 x 2 weeks. Throughout weeks 2-5 and 7-10.
  Total energy expenditure measured by DLW for the 4 week BB and BD diet phases
Resting Metabolic Rate (RMR) | Baseline,week 1, week 5, week 6, week 10.
  RMR measured with indirect calorimetry (ventilated hood)
Thermic effect of food (TEF) | Week 1, week 5, week 6, week 10.
  TEF measured with indirect calorimetry (ventilated hood) for 6 hours after a breakfast meal
Body Volume | Week 1, week 5, week 6, week 10.
  Measured with Air Displacement plethysmography (BODPOD),
Bone Mineral Content | Week 1, week 5, week 6, week 10.
  Measured with Dual energy x-ray absorptiometry (DEXA)
Total Body Water | Week 1, week 5, week 6, week 10.
  Measured with deuterium dilution
Body Composition | Week 1, week 5, week 6, week 10.
  4 compartment model to assess changes in body composition (Combined from the measures of body weight, body volume, total body water and bone mineral)
Gastric emptying | Week 1, week 5, week 6, week 10.
  Gastric emptying measured using stable isotope, Octanoic acid labelled breath samples.
Waist and hip circumference | Week 1, week 5, week 6, week 10.
  Change in waist and hip circumferences and waist to hip ratio
Gut appetite hormones | Week 1, week 5, week 6, week 10.
  Change in plasma fasting and 2 hr post-meal appetite hormones
Plasma glucose | Week 1, week 5, week 6, week 10.
  Change in plasma fasting and 2 hr post-meal glucose
Plasma insulin | Week 1, week 5, week 6, week 10.
  Change in plasma fasting and 2 hr post-meal insulin
Blood lipids | Week 1, week 5, week 6, week 10.
  Change in plasma fasting and 2 hr post-meal blood lipids
Daily Subjective Appetite | Hourly measures for 3 days in week 1,week 5, week 6, week 10.
  Changes in subjective appetite (hunger, fullness, desire to eat) measured using visual analogue scale questionnaires every waking hour for 3 days.
Postprandial Subjective Appetite | Week 1, week 5, week 6, week 10.
  Changes in subjective appetite (hunger, fullness, desire to eat) measured using visual analogue scale questionnaires every 30 minutes for 6 hours after test meals.
Faecal sample analysis for gut health | Week 1, week 5, week 6, week 10.
  Chronic influence on changes in gut microbiota
Physical activity | Measured continuously for 24 hours for 3 days in week 1,week 5, week 6, week 10.
  Change in physical activity levels measured with accelerometer (actigraph)
24 hour blood glucose | Measured continuously for 24 hours for 3 days in week 1,week 5, week 6, week 10.
  Changes in 24 hour blood glucose levels measured with a continuous glucose monitor

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra M Johnstone, PhD, Principal Investigator — University of Aberdeen
Locations (1):
- The Rowett Institute, Aberdeen, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ruddick-Collins LC, Morgan PJ, Fyfe CL, Filipe JAN, Horgan GW, Westerterp KR, Johnston JD, Johnstone AM. Timing of daily calorie loading affects appetite and hunger responses without changes in energy metabolism in healthy subjects with obesity. Cell Metab. 2022 Oct 4;34(10):1472-1485.e6. doi: 10.1016/j.cmet.2022.08.001. Epub 2022 Sep 9. PMID 36087576